CLINICAL TRIAL: NCT06602310
Title: Evaluation of the Utility of the Preanestes@s2.0, a Web Based Application for Preoperative Assessment. Comparison of the Rate of Suboptimal Web Based Telematic Assessments Versus the Outpatient Visit.
Brief Title: Utility of Preanestes@s2.0, a Web Based Application for Preoperative Assessment.
Acronym: Preanestes@s
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has been terminated due to technical limitations in the institutional IT system, which cannot support the maintenance and integration of the application. Consequently, no further participant recruitment will be conducted.
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PREANEST.2.0
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Mobile Application; Preoperative Period; Internet-based Intervention; Surgical Procedures, Elective; Assessment Evaluation
Keywords: Electronic Health Records; Health Impact Assessment; Patient Health Questionnaire; Preoperative Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preanestes@s2.0: web-based non-face-to-face preoperative assessment. Telematic group. (Experimental): Participants will be leaded through preoperative period on a web based application. Participants will be addressed to either virtual or telephone POA on the basis of the information registered in the web based preoperative questionnaire that the application incorporates. Virtual assessment will be performed by evaluating both the filled web based questionnaire together with participants´ electronic medical records. Telephone assessment will also incorporate a telephone call for further clarifications.
  Interventions: Other: Web based preoperative assessment
- Traditional face-to-face preoperative assessment (No Intervention): Participants will be leaded through preoperative period following traditional institutional standards of care. Face to face assessment will be performed in the traditional way by means of an interview with the participant together with the consultation of participant´s previous electronic records.

INTERVENTIONS:
Other: Web based preoperative assessment — Preoperative assessment conducted through a web based application. Telematic non-face-to-face preoperative assessment.
  Arms: Preanestes@s2.0: web-based non-face-to-face preoperative assessment. Telematic group.

SUMMARY:
The use of web based self-assessment questionnaires as a complementary tool for conducting preoperative assessment (POA) is gaining increasing acceptance. Preanestes@s2.0 is a web based application fully developed by the investigators team which potentially allows for remote non-telephonic POA. It has already been evaluated as a feasible tool in terms of patient acceptance and quality of the information recorded. In this prospective two-arm study, the investigators will evaluate the incidence of suboptimal POA when the participants are evaluated through Preanestes@s2.0 versus the traditional outpatient face to face visit. The investigators will consider as suboptimal any POA that potentially may generate an inadequate preparation of the patient which may affect the expected results. A total 1.127 participants will be evaluated through Preanestes@s2.0 (intervention arm) and compared to a cohort of 1.127 patients evaluated by traditional face-to-face interview (non-intervention arm). The comparison will be made by means of a propensity score matching study. Patients included in both arms of the study will be recruited throughout the same period of time.

DETAILED DESCRIPTION:
Preoperative evaluation models that integrate the use of electronic health records and telephone or electronic questionnaires are evolving aiming to optimize the preoperative assessment process. In 2018, the investigators developed Preanestes@s, a web based application conceived to allow for remote preoperative assessment and guide patients through the preoperative period. The application includes a patient interface which offers general and individualized information on the preoperative process, with the possibility of generating a dynamic interaction between patients and medical staff. Patient interface incorporates a smart web based preoperative questionnaire (PreQuest), which once fully completed automatically classifies patients as per their American ASA grade (from the American Society of Anesthesia Physical Status Classification), and suggests the convenience of a face-to-face visit (f-visit) versus a virtual non-face-to-face non-telephonic visit (v-visit) according to the assigned ASA grade (patients with ASA grade≥3 are systematically recommended for f-visit) and the presence of predefined comorbidities or physical conditions not necessarily related to a specific ASA grade (i.e., current or persistent cough or dyspnea). Both virtual and f-visit are performed by an anesthesiologist. Preanestes@s also determines the preoperative tests that should be conducted according to the patient's condition and offers individualized health advice and recommendations on treatment, with the option of electronically signing an experimental model of electronic informed consent.

In its original version, Preanestes@s has been evaluated both in terms of user acceptance and usability, as well as in terms of the quality of information recording, this last by means of a paired study which compared the information recorded through PreQuest with that recorded by the anesthesiologist when performing the v-visit and the f-visit. The results have been favorable to the model, both in terms of user acceptance and of the quality of the information recording.

On april 2021 the investigators launched a prospective study to evaluate the feasibility and utility of the model, this estimated by comparing the rate of suboptimal preoperative studies carried out using the application versus the traditional outpatient f-visit (Evaluation of the Utility of Preanestes@s, a Web Based Application for Preoperative Assessment; NCT04787783). Unfortunately, the study recruitment rate has been lower than expected, partly due to the difficulties derived from the limited collaboration of the surgeons, the actors initially proposed to lead the recruiting process (recruitment should preferably take place at the time of the surgical indication at the surgeon´s office). Once the investigators detected the difficulties in recruiting by surgeons, they considered filling this shortage through the figure of a recruiting agent, but the investigators were forced to discontinue this task due to lack of funding, what finally led them to seek alternatives to improve the effectiveness and efficiency of the model. From that moment on, the investigators began to work with the objective of achieving automatic patient recruitment. This is how the Preanestes@s2.0 version came about.

Preanestes@s2.0 incorporates a new automatic recruitment interface, so that information that previously had to be entered by the surgeon or, in its defect, by a recruiting agent, is now filled in automatically. Similarly, the new patient management interface has also been improved in automatism and simplified, so that the information that previously had to be managed by the administrative staff is now managed automatically.

On the other hand, the f-visit has been replaced by a telephone visit (t-visit), so that the options available in the model would be the v-visit (non face-to-face non-telephone) and the t-visit (non face-to-face but telephone), regardless of the fact that the anesthesiologist evaluating each case may request a f-visit on demand for specific cases.

Preanestes@s2.0 also automates the patient appointment process, thus reducing the administrative workload and improving the efficiency of the model.

Finally, Preanestes@s2.0 also improves its capabilities when communicating with the patient, with the incorporation, among others, of WhatsApp messaging.

Assuming the improvements of the model and taking into account that they represent a relevant modification to the conditions of the original study, the investigators designed a new prospective work aimed at comparing the rate of adequate preoperative assessments using the Preanestesas2.0 application versus the traditional face-to-face model.

This study (Internal code SICEIA-2024-001682) has been approved by the local Ethics Committee -Comité de Ética e Investigación de los Hospitales Universitarios Virgen Macarena y Virgen del Rocío-and signed by its Secretary José Carlos García Pérez, date 26.07.2024.

In this study, the objective of the investigators is to assess whether the use of a web based application for the preoperative assessment allows an adequate completion of the preoperative process when compared to traditional face-to-face outpatient interview. The quality of the information recorded by this web based application has been previously tested by the investigators showing promising results in terms of security and accuracy.

The investigators have designed a prospective two-arm study to compare the performance of the two modalities of preoperative assessment: web based versus face to face outpatient visit.

The investigators will base their evaluation of performance on previously published criteria: the Andalusian Regional Government Health Council defines a suboptimal preoperative assessment (SOPA) as one that potentially generates an inadequate preparation of the patient that may affect the expected results. Specific criteria defining SOPA are detailed in the Outcomes Measures section of the present document.

A total 1.127 participants will be evaluated through Preanestes@s2.0 (Intervention arm) and compared to a cohort of 1.127 patients evaluated by traditional face-to-face interview (Non-intervention arm).

Allocation of participants to Intervention arm will be consecutive and based on daily distribution of the clinics: Orthopedics, General Surgery and Urology. Participants in the Non-intervention group will be recruited ex-post, using the propensity score methodology among patients assessed by the traditional face to face format throughout the study period.Written informed consent will be obtained of all participants in the Intervention group prior to their recruitment.

Statistical analysis Data collection and subsequent analysis will be performed by the investigators team. Qualitative variables will be represented through the absolute and marginal frequencies. The investigators will analyze the incidence of SOPA in both groups, using Chi square to study the difference between the proportions in the case of normal distribution, or, failing that, the Mann-Whitney U. In the same way, the investigators will study the differences for each of the defining criteria of SOPA.

Sample Siz: following the model of Kinley et al in the study comparing the quality of the pre-anesthesia record carried out by anesthesia trainees versus trained nurses, the investigators will use the variable Incomplete studies that could have affected perioperative management for the calculation of the sample size. This variable would be equivalent to the variable SOPA in present work. Based on Kinley data, the investigators will use an incomplete study rate of 15%, a figure that coincides with the standard Inadequate assessment in the Guide for the Perioperative Process published by the Andalusian Regional Government Health Council, which establishes a maximum; acceptable; rate of inadequate completion of the preoperative protocols in 15%. In this study of equivalence between the two formats, the investigators will assume equivalence if a maximum difference of 25% between both formats is observed, which represents a differential of 3.75% over the initial 15%. Thus, for a two-sided calculation and assuming an alpha error of 0.05 and a beta error of 0.2 (80% power), it would be necessary to include 1,127 participants per group.

ELIGIBILITY:
Inclusion Criteria:

* Participants undergoing day scheduled surgery in our institutions: Hospitales Universitarios Virgen del Rocío y Virgen Macarena.
* Surgical specialities included: Urology, General Surgery, Orthopedics, Ear, nose, and throat surgery.

Exclusion Criteria:

* Urgent procedures, oncologic procedures, patients without the ability to understand informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2254 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Suboptimal preoperative assessments (SOPA). | From the day of intervention up to 7 days after intervention
  Dichotomous (present/absent) composite variable comprising any of the following:
  1. Lack of relevant information in the preoperative assessment that conducts to: - Inadequate conciliation of chronic medication - Inadequate preoperative fasting - Inadequate register of clinical or functional conditions that may cause delayed intervention the day of surgery (presence of uncontrolled chronic diseases, presence of impaired functional status undetected in the preoperative assessment, etcetera.
  2. Lack of complementary tests indicated according to preoperative protocol
  3. Presence of not indicated complementary tests according to preoperative protocol
  4. Lack of properly filled informed consent
  5. Cancellation of the intervention due to inadequate preoperative preparation (attributable to mismanagement of preoperative information)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen Del Rocío, Seville

REFERENCES:
- [Result] Goodhart IM, Andrzejowski JC, Jones GL, Berthoud M, Dennis A, Mills GH, Radley SC. Patient-completed, preoperative web-based anaesthetic assessment questionnaire (electronic Personal Assessment Questionnaire PreOperative): Development and validation. Eur J Anaesthesiol. 2017 Apr;34(4):221-228. doi: 10.1097/EJA.0000000000000545. PMID 27798453
- [Result] Arias A, Benitez S, Canosa D, Borbolla D, Staccia G, Plazzotta F, Casais M, Michelangelo H, Luna D, Bernaldo de Quiros FG. Computerization of a preanesthetic evaluation and user satisfaction evaluation. Stud Health Technol Inform. 2010;160(Pt 2):1197-201. PMID 20841873
- [Result] Zaballos M, Lopez-Alvarez S, Argente P, Lopez A; Grupo de Trabajo de Pruebas Preoperatorias. Preoperative tests recommendations in adult patients for ambulatory surgery. Rev Esp Anestesiol Reanim. 2015 Jan;62(1):29-41. doi: 10.1016/j.redar.2014.07.007. Epub 2014 Aug 18. English, Spanish. PMID 25146773
- [Result] De Hert S, Staender S, Fritsch G, Hinkelbein J, Afshari A, Bettelli G, Bock M, Chew MS, Coburn M, De Robertis E, Drinhaus H, Feldheiser A, Geldner G, Lahner D, Macas A, Neuhaus C, Rauch S, Santos-Ampuero MA, Solca M, Tanha N, Traskaite V, Wagner G, Wappler F. Pre-operative evaluation of adults undergoing elective noncardiac surgery: Updated guideline from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2018 Jun;35(6):407-465. doi: 10.1097/EJA.0000000000000817. PMID 29708905
- [Result] Kinley H, Czoski-Murray C, George S, McCabe C, Primrose J, Reilly C, Wood R, Nicolson P, Healy C, Read S, Norman J, Janke E, Alhameed H, Fernandes N, Thomas E. Effectiveness of appropriately trained nurses in preoperative assessment: randomised controlled equivalence/non-inferiority trial. BMJ. 2002 Dec 7;325(7376):1323. doi: 10.1136/bmj.325.7376.1323. PMID 12468478
- [Result] Conde JM, Moreno-Conde A, Salas-Fernandez S, Parra-Calderon CL. ITCBio, a Clinical and Translational Research Platform. AMIA Annu Symp Proc. 2020 Mar 4;2019:673-680. eCollection 2019. PMID 32308862
- [Result] Lozada MJ, Nguyen JT, Abouleish A, Prough D, Przkora R. Patient preference for the pre-anesthesia evaluation: Telephone versus in-office assessment. J Clin Anesth. 2016 Jun;31:145-8. doi: 10.1016/j.jclinane.2015.12.040. Epub 2016 Apr 15. PMID 27185698
- [Result] Law TT, Suen DT, Tam YF, Cho SY, Chung HP, Kwong A, Yuen WK. Telephone pre-anaesthesia assessment for ambulatory breast surgery. Hong Kong Med J. 2009 Jun;15(3):179-82. PMID 19494372
- [Result] Ludbrook G, Seglenieks R, Osborn S, Grant C. A call centre and extended checklist for pre-screening elective surgical patients - a pilot study. BMC Anesthesiol. 2015 May 19;15:77. doi: 10.1186/s12871-015-0057-1. PMID 25985775
- [Result] Blanco Vargas D, Faura Messa A, Izquierdo Tugas E, Santa-Olalla Bergua M, Noguera Sopena MM, Manoso Noriego M. [Online versus non-standard face to face preoperative assessment: cost effectiveness]. Rev Esp Anestesiol Reanim. 2012 Aug-Sep;59(7):350-6. doi: 10.1016/j.redar.2012.05.039. Epub 2012 Jul 10. Spanish. PMID 22784647
- [Result] Applegate RL 2nd, Gildea B, Patchin R, Rook JL, Wolford B, Nyirady J, Dawes TA, Faltys J, Ramsingh DS, Stier G. Telemedicine pre-anesthesia evaluation: a randomized pilot trial. Telemed J E Health. 2013 Mar;19(3):211-6. doi: 10.1089/tmj.2012.0132. Epub 2013 Feb 5. PMID 23384334
- [Result] de la Matta M, Alonso-Gonzalez M, Moreno-Conde J, Salas-Fernandez S, Lopez-Romero JL; Preanestesas study investigators. Development and patient acceptance of Preanestes@s, a web-based application and electronic questionnaire for preoperative assessment. A prospective cohort study. Rev Esp Anestesiol Reanim (Engl Ed). 2022 Aug-Sep;69(7):383-392. doi: 10.1016/j.redare.2022.01.002. Epub 2022 Jul 20. PMID 35871145
- [Result] de la Matta M, Alonso-Gonzalez M, Garcia-Santigosa M, Arance-Garcia M, Sanchez-Pena J, Castro-Linan LM, Lopez-Romero JL. Accuracy and Comprehensiveness in Recording Information of a Web-Based Application for Preoperative Assessment: A Prospective Observational Study. J Perianesth Nurs. 2023 Jun;38(3):440-447. doi: 10.1016/j.jopan.2022.08.004. Epub 2022 Dec 9. PMID 36509667